CLINICAL TRIAL: NCT05224401
Title: Pivmecillinam With Amoxicillin/Clavulanic Acid for Step Down Oral Therapy in Febrile UTIs Caused by ESBL-producing Enterobacterales (PACUTI)
Brief Title: Pivmecillinam With Amoxicillin/Clavulanic Acid for Step Down Oral Therapy in ESBL UTIs
Acronym: PACUTI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-PACUTI
Record Dates: First submitted 2021-12-14; First posted 2022-02-04 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Urinary Tract Infections; Bacteremia; Antibiotic Resistant Infection
MeSH Terms: conditions — Urinary Tract Infections; Bacteremia | interventions — Amdinocillin Pivoxil; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin; Trimethoprim; Sulfamethoxazole; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PAC treatment (Experimental)
  Interventions: Drug: Pivmecillinam and amoxicillin/clavulanic acid
- Standard treatment (Active Comparator)
  Interventions: Drug: Standard treatment, ciprofloxacin, trimethoprim/sulfamethoxazole or ertapenem depending on susceptibility

INTERVENTIONS:
Drug: Pivmecillinam and amoxicillin/clavulanic acid — 1 tablet pivmecillinam 400 mg and 1 tablet Amoxicillin/clavulanic acid 875/125 mg, three times daily.
  Other Names: Coactin or selexid etc, and Augmentin or Clavulin etc
  Arms: PAC treatment
Drug: Standard treatment, ciprofloxacin, trimethoprim/sulfamethoxazole or ertapenem depending on susceptibility — Ciprofloxacin 500 mg twice daily, trimethoprim/sulfamethoxazole 800 mg/160 mg twice daily or ertapenem 1 g once daily.
  Other Names: Bactrim
  Arms: Standard treatment

SUMMARY:
To evaluate if the combination of pivmecillinam and clavulanic acid (PAC) is non-inferior to ciprofloxacin, trimethoprim-sulfamethoxazole or ertapenem as step down oral therapy in patients with febrile UTI caused by extended spectrum beta-lactamase (ESBL) producing Enterobacterales (EPE).

DETAILED DESCRIPTION:
A recent observational cohort study supports the notion that beta-lactams can be used with similar efficacy to fluoroquinolones as step down therapy in bacteremic E. coli UTI's. As such, pivmecillinam clavulanic acid (PAC) constitute an appealing per oral alternative, but the combination's safety and efficacy has not been evaluated in a clinical trial The aim of this trial is to investigate whether the PAC combination is non-inferior to ciprofloxacin, trimethoprim-sulfamethoxazole or ertapenem as step down oral therapy in treating EPE-causing febrile UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Fever (≥ 38.3 C) or shaking chills at least once at home or in hospital
3. Clinical suspicion of UTI including at least one of the following symptoms:

   1. Dysuria, urinary urgency, difficulty urinating, new or worsened urinary incontinence, macroscopic haematuria or increased urinary frequency
   2. Low abdominal pain or flank pain with percussion or palpation tenderness over kidneys and/or bladder.
4. Urine (≥ 103 CFU/mL) and/or blood culture positive for EPE* with susceptibility to pivmecillinam†.
5. In-patient who has received 1-5 days of EPE-active‡ intravenous antibiotics
6. Discontinuing parenteral treatment and starting treatment with oral antibiotics is considered safe according to the treating physician.

   * EPE refers to ESBL-producing Enterobacterales. This includes Escherichia coli, Klebsiella pneumoniae, Proteus mirabilis, Klebsiella oxytoca, and Citrobacter koseri.

     * Susceptibility for pivmecillinam in the study is based on zone diameter breakpoints for pyelonephritis (≥ 20 mm) which was received by personal communication with professor Christian Giske, the chairman of the European Committee of Antimicrobial Susceptibility Testing (EUCAST) (26).

       * EPE-active intravenous antibiotics refers to EUCAST susceptibility testing and will most often be piperacillin-tazobactam, meropenem or imipenem-cilastatin in the Swedish setting, and less often aminoglycosides or newer beta-lactamase-inhibitor-containing beta-lactam antibiotics (27). Participants who have only received one dose of EPE-active intravenous antibiotics are also eligible and are considered within the "1-5 days" of antibiotics.

Patients may only be recruited and randomised once in this trial.

Exclusion criteria (any of the following)

1. Known or suspected pregnancy.
2. Known or suspected life-threatening allergy towards beta-lactam antibiotics.
3. Clinical isolate of EPE is resistant to ciprofloxacin, TMX and ertapenem.
4. Severe renal insufficiency with estimated glomerular filtration rate (eGFR) <10mL/min or requiring any form of dialysis.
5. Severe decompensated liver failure (i.e., child Pugh class B or C).
6. Genetic metabolic diseases associated with severe carnitine deficiency.
7. Megaloblastic haematopoiesis.
8. Co-treatment with valproate or valproic acid (due to interaction with pivmecillinam and ertapenem respectively)
9. Other reason to which patient is unfit to be included in the study according to treating physician, e.g., cognitive impairment preventing informed consent and follow-up, inability to speak and/or read Swedish, missing national personal identification number or missing telephone number preventing follow-up or planned duration of antibiotics > 10 days due to complicating factors.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | Clinical cure 10 days (+/- 2 days)
  Clinical cure defined as being alive with absence of fever (≥ 38.3 C) and resolution of, or return to non-infected baseline of, urinary tract symptoms (as defined in inclusion criteria) without additional antibiotic treatment (for UTI symptoms) based on fever control and a semi-structured interview at a live return visit to an independent physician (i.e. not previously involved in the care of the study participant) at an infectious disease clinic.

SECONDARY OUTCOMES:
To compare the recurrence prevalence of EPE (phenotypically same species) in urine cultures 10 +/- 2 days after antibiotic treatment between groups (i.e., microbiological cure). | Up to 28 days
  Yes or no.
To compare the prevalence of EPE or carbapenemase-producing bacteria in faecal cultures 10 +/- 2 days after antibiotic treatment between groups. | Up to 28 days
  Yes or no.
To compare participants' perception of treatment tolerability | 10 days
  Tolerability is measured on a 1-10 scale.
To compare the incidence of early study drug discontinuation between groups. | 10 days
  Yes or no.
To compare the incidence of additional antibiotic subscriptions (for UTI) within 28 days between groups. | 28 days
  Yes or no.
To compare re-admission to hospital (due to UTI-related symptoms) within 28 days between groups. | 28 days
  Yes or no.
To compare the incidence of drug-related serious adverse events (SAE) within 28 days between groups. | 28 days
  Yes or no.
To compare the all-cause mortality within 28 days between groups. | 28 days
  Yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ljungquist, MD, PhD., Principal Investigator — Lunds universitet; Emeli Månsson, MD, PhD., Study Chair — Västmanland Hospital Västeras
Locations (5):
- Sweden (5):
  - Helsingborg hospital, Helsingborg
  - Kristianstad hospital, Kristianstad
  - Skåne University Hospital, Lund, Lund
  - Skåne University Hospital, Malmö, Malmo
  - Västmanland hospital Västerås, Västerås

IPD SHARING:
Plan to Share IPD: Undecided
Yes.

REFERENCES:
- [Background] Saad S, Mina N, Lee C, Afra K. Oral beta-lactam step down in bacteremic E. coli urinary tract infections. BMC Infect Dis. 2020 Oct 21;20(1):785. doi: 10.1186/s12879-020-05498-2. PMID 33087051
- [Derived] Tverring J, Mansson E, Andrews V, Ljungquist O. Pivmecillinam with Amoxicillin/Clavulanic acid as step down oral therapy in febrile Urinary Tract Infections caused by ESBL-producing Enterobacterales (PACUTI). Trials. 2023 Sep 2;24(1):568. doi: 10.1186/s13063-023-07542-3. PMID 37660037